CLINICAL TRIAL: NCT04498689
Title: A Phase II, Single-arm Study to Evaluate the Efficacy and Safety of PD-1 Antibody Camrelizumab in Combination With Nab-paclitaxel Plus Gemcitabine in Treating Patients With Metastatic Pancreatic Cancer
Brief Title: Efficacy and Safety of Camrelizumab Combined With Nab-Paclitaxel Plus Gemcitabine for Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Vice President, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-27
Record Dates: First submitted 2020-06-30; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Metastatic pancreatic cancer; Pancreatic Adenocarcinoma; Camrelizumab; Nab-paclitaxel; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — camrelizumab; Taxes; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- camrelizumab + nab-paclitaxel + gemcitabine (Experimental): PD-1 Monoclonal Antibody Camrelizumab at 200 mg on Day 1 and 15 nab-paclitaxel at 100 mg/m2 on Day 1, 8, and 15; gemcitabine at 1000 mg/m2 on Day 1, 8, and 15
  Interventions: Drug: Camrelizumab; Drug: Nab paclitaxel; Drug: Gemcitabine Injection

INTERVENTIONS:
Drug: Camrelizumab — Patients firstly receive camrelizumab 200 mg per time (iv, no less than 20 minutes and no more than 60 minutes, rinse time included) on Day 1 and 15 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks until the disease recurrence, unacceptable toxicity, death or begin a novel therapeutic.
Drug: Nab paclitaxel — Patients secondly receive nab-paclitaxel 100 mg/m2 (iv, at least 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks until the disease recurrence, unacceptable toxicity, death or begin a novel therapeutic.
  Other Names: Albumin paclitaxl
Drug: Gemcitabine Injection — At last, patients receive gemcitabine 1000 mg/m2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment. Treatment repeats every 4 weeks until the disease recurrence, unacceptable toxicity, death or begin a novel therapeutic.
  Other Names: Gemcitabine

SUMMARY:
The present study is intended to investigate the objective response rate (ORR) and the progression-free survival (PFS) of the patients with histologically- or cytologically-confirmed metastatic pancreatic cancer after treating with the combination of camrelizumab, gemcitabine and nab-paclitaxel, and to investigate the overall survival (OS) and the adverse event (AE) of the patients with histologically- or cytologically-confirmed metastatic pancreatic cancer after treating with the combination of camrelizumab, gemcitabine and nab-paclitaxel.

DETAILED DESCRIPTION:
This a prospective, single-arm, open-label, phase 2 studye evaluating the efficacy and safety of camrelizumab, gemcitabine and nab-paclitaxel for metastatic pancreatic cancer patients. The primary endpoints are ORR and PFS, and the secondary are OS and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed informed consent form obtained prior to treatment. The patients were fully explained and understood the purpose, contents, predicted efficacy, pharmacological effects, and risks of this study.

  2. target patients
  1. the patients were histopathologically- or cytocologically-confirmed as metastatic pancreatic cancer.
  2. At least one measurable objective lesion (both primary and metastatic) was identified based on the RECIST 1.1 criteria;
  3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
  4. The expected survival after surgery ≥ 3 months
  5. The subjects have good compliance, can be treated and followed up, and voluntarily comply with the relevant provisions of this study
  6. No contraindications for camrelizumab, gemcitabine and nab-paclitaxel. 3. Age and reproductive status

  <!-- -->

  1. Male and female patients at the age of 18-75
  2. Subjects of child-bearing age must agree to take effective contraceptive measures during the study period; Serum or urine pregnancy tests must be negative for women of childbearing age 24 hours before the start of therapy;
  3. Women must not lactate.

     Exclusion Criteria:
* 1. The target disease has cerebral metastasis; 2. Previously treated by anti-PD-1 or anti-PD-L1 drugs; 3. Received any investigational drug within 4 weeks before the first use of the research drug; 4. Enrolled in another clinical study, unless it is an observational (non-interventional) clinical study or an interventional follow-up clinical study; 5. medical history and complications

  1. patients had uncontrolled serious medical condition that the investigator considered may affect the subject's to receive treatment under the study program. For example, patients with severe medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc.
  2. patients who are suffering active, known or suspected autoimmune diseases (including but limited to uveitis, enteritis, hepatitis, pituitary inflammation, nephritis, vasculitis, hyperthyroidism, hypothyroidism and asthma requiring bronchodilator therapy, etc.). Subjects with hypothyroidism who only need hormone replacement therapy and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, or hair loss) can be enrolled;
  3. Patients who are suffering from active tuberculosis infection: Patients with active pulmonary tuberculosis infection within 1 year before medication should be excluded even if they have been treated; patients with a history of active tuberculosis infection more than 1 year ago should also be excluded unless it is proven that they have received standard anti-TB treatment before;
  4. Patients who have previous interstitial lung disease or (non-infectious) pneumonia and requires oral or intravenous steroid therapy;
  5. Patients who need to receive long-term systemic hormones (dose equivalent to >10mg prednisone/day) or any other form of immunosuppressive therapy. Subjects using inhaled or topical corticosteroids can be enrolled;
  6. Patients who have uncontrolled heart disease, such as:

     1. New York Heart Association (NYHA) level 2 heart failure;
     2. Unstable angina;
     3. Myocardial infarction occurred within 1 year
     4. Supraventricular or ventricular arrhythmias that have clinical significance and require treatment or intervention
  7. Dementia, changing of mental state or any mental illness which could hinder understanding or informed consent or fill out questionnaires;
  8. History of allergy or hypersensitivity to any therapeutic ingredient;
  9. Combined with other malignant tumors excepted pancreatic cancer within the first 5 years of randomization, excepted well-treated basal cell or squamous cell carcinoma of the skin, localized prostate cancer after radical resection, and ductal carcinoma in situ of the breast after radical resection;
  10. Previously received systemic therapy for advanced/metastatic pancreatic cancer;
  11. Subjects who had previously been pathologically diagnosed with squamous cell carcinoma (no organ limitation) and received neoadjuvant/adjuvant therapy with taxa regimen.
  12. Patients who had Grade 2 or above Peripheral neuropathy according to CTCAE Ver. 5.0.

  6. Abnormal results of physical examination and laboratory examination
  1. Absolute neutrophil count (ANC) ≥ 1.5×109/L; Platelets (PLT) ≥ 80×109/L; Hemoglobin (Hb) ≥ 90g/L
  2. Aspartate aminotransferase (AST, or serum glutamic oxaloacetic transaminase, SGOT) and alanine aminotransferase (ALT, or serum glutamic pyruvate transaminase, SGPT) > 2.5 × ULN (institutional upper limit of normal), > 5 ×ULN (hepatic metastases occasion); Total bilirubin (TBIL)>1.5 × ULN;
  3. Creatinine (CRE)> 1.5 × ULN
  4. Prothrombin time (PT) and international normalized ratio (INR) > 1.5 × ULN. Or activated partial thromboplastin time (aPTT) > 1.5 × ULN. Unless the subject had received anticoagulant treatment
  5. Subjects had hepatitis b surface antigen (HBsAg)-positive and HBV-DNA titer in peripheral blood greater than or equal to 1000 copy number /L; If HBsAg is positive and the HBV-DNA of peripheral blood ≥ 1000 copy number/L, the subjects will be eligible for inclusion if the investigator considers that chronic hepatitis b is stable and does not increase the risk of subjects.

  4. Human immunodeficiency virus (HIV)- or hepatitis C virus (HCV) positive patients; 5. Patients who suffer from active infection requiring systemic treatment; 6. Patients need other concomitant anti-tumor drugs; 7. Participation in any trial drug treatment or another interventional clinical trial 30 days before screening period.

  8. Other conditions that the investigators considered are not suitable for the enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | from enrollment to time of evaluation or date of death from any cause, whichever came first, estimated 18 months
  To evaluate the Overall Response Rate of patients with metastatic pancreatic cancer after the treatment of camrelizumab with nab-paclitaxel plus gemcitabine.
Progression Free Survival | from enrollment to time of evaluation or date of death from any cause, whichever came first, estimated 18 months
  To evaluate the Progression Free Survival of patients with metastatic pancreatic cancer after the treatment of camrelizumab with nab-paclitaxel plus gemcitabine.

SECONDARY OUTCOMES:
overall survival | from enrollment to time of evaluation or date of death from any cause, whichever came first, estimated 18 months
  To evaluate the overall survival of patients with metastatic pancreatic cancer after the treatment of camrelizumab with nab-paclitaxel plus gemcitabine.
adverse events | from enrollment to time of evaluation or date of death from any cause, whichever came first, estimated 18 months
  To evaluate the adverse events of patients with metastatic pancreatic cancer after the treatment of camrelizumab with nab-paclitaxel plus gemcitabine.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Yu, Principal Investigator — Fudan University
Locations (1):
- Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No